CLINICAL TRIAL: NCT01474772
Title: A Phase 3b Multicenter, Double-blind, Randomized, Placebo-controlled Cross-over Efficacy And Safety Study Of Pregabalin In The Treatment Of Patients With Painful Diabetic Peripheral Neuropathy And Pain On Walking
Brief Title: Efficacy and Safety Study of Pregabalin in the Treatment of Pain on Walking in Patients With Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0081269; 2011-003266-32 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2014-11

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Pain on Walking; Pregabalin
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabain (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Pregabalin — 150-300 mg/day given in 3 divided doses as capsules
  Other Names: Lyrica
  Arms: Pregabain
Other: placebo — matching placebo capsules given in 3 divided doses
  Arms: Placebo

SUMMARY:
The intent of this study is to treat subjects with painful Diabetic Peripheral Neuropathy (DPN) who also have pain on walking and to determine whether or not pregabalin demonstrates improvement relative to placebo on the following: reducing DPN pain, reducing pain on walking, and providing other benefits associated with daily activities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are at least 18 years old.
* Diagnosis of painful diabetic peripheral neuropathy.
* Pain on walking.

Exclusion Criteria:

* Inability to walk 50 feet on a flat surface.
* Pain on walking due to conditions other than diabetic peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (34):
  - Dedicated Clinical Research, Goodyear, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - HealthCare Partners Medical Group, Los Angeles, California
  - IDS Pharmacy, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - PAB Clinical Research, Brandon, Florida
  - Pulmonary Associates of Brandon, Brandon, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - The Office of Laszlo Jozef Mate, MD, North Palm Beach, Florida
  - Meridien Research, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Columbus Research Foundation, Columbus, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - The Office of Dr. Stephen H. Miller, MD, Las Vegas, Nevada
  - The Medical Research Network, LLC, New York, New York
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - The Office of Veronique Sebastian, MD, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Health and Science University - Comprehensive Pain Center, Portland, Oregon
  - Oregon Health and Science University - Department of Anesthesiology and Perioperative Medicine, Portland, Oregon
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Neurology and Pain Clinic, LLC, Orangeburg, South Carolina
  - Houston Neurocare, Houston, Texas
  - Centex Research, Inc., Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
- Czechia (3):
  - Privatni specializovana ambulance pro neurologii a detskou neurologii, Brno-Bystrc
  - Clintrial, s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
- South Africa (4):
  - Dr DR Lakha's Practice, Johannesburg, Gauteng
  - Dr Hemant Makan (Private Practice), Lenasia, Gauteng
  - Randles Road Medical Centre, Durban, KwaZulu-Natal
  - Richards Bay Trial Centre, Richards Bay
- Sweden (4):
  - Forskningsmottagningen Gamla Sjukhuset i Falkoping, Falköping
  - Center for Lakemedelsstudier, Malmo
  - Citydiabetes, Stockholm
  - Bragee Medect AB, Stockholm

REFERENCES:
- [Derived] Huffman C, Stacey BR, Tuchman M, Burbridge C, Li C, Parsons B, Pauer L, Scavone JM, Behar R, Yurkewicz L. Efficacy and Safety of Pregabalin in the Treatment of Patients With Painful Diabetic Peripheral Neuropathy and Pain on Walking. Clin J Pain. 2015 Nov;31(11):946-58. doi: 10.1097/AJP.0000000000000198. PMID 25565583
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081269&StudyName=Efficacy%20and%20Safety%20Study%20of%20Pregabalin%20in%20the%20Treatment%20of%20Pain%20on%20Walking%20in%20Patients%20with%20Diabetic%20Peripheral%20Neuropathy%20%28DPN%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 411 participants were screened, of whom 206 were withdrawn before randomization. 205 were randomized, of whom 2 discontinued before being treated. Participants were randomized at 36 centers in 4 countries: US (25), Sweden (4), South Africa (4), and Czech Republic (3). 11 centers received study drug but did not randomize participants.
Pre-assignment Details: Participants completed daily pain and sleep diary from Visit 1 (V1; Screening) to Visit 12 (V12; Follow-up). Participants with a mean pain score ≥ 4 (moderate to severe pain) and those meeting the pain on walking criteria (post-walk pain score ≥ 4, and > the pre-walk pain score at V1 and Visit 2 [V2; Baseline]) were randomized.
Groups:
- Pregabalin/Placebo: Participants were randomized to double-blind treatment with pregabalin for 6 weeks (2 week dose titration [starting dose: 150 mg/day] and 4 weeks fixed dose [150 - 300 mg/day]) in period 1 followed by placebo in period 2. There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
- Placebo/Pregablin: Participants were randomized to double-blind treatment with placebo for 6 weeks in period 1 followed by pregabalin in period 2 (2 week dose titration [starting dose: 150 mg/day] and 4 weeks fixed dose [150 - 300 mg/day]). There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
Period: Period 1
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 101 (STARTED=treated. In Period 1 a participant discontinued due to an AE and later died due to the AE.) | 102 (STARTED=treated)
Completed | 89 | 99
Not Completed | 12 | 3
Not completed — Adverse Event (AE) Related to Study Drug | 6 | 1
Not completed — AE not Related to Study Drug | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Reason not Specified | 1 | 1
Period: Washout
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 89 | 99
Completed | 86 | 97
Not Completed | 3 | 2
Not completed — AE not Related to Study Drug | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Reason not Specified | 0 | 1
Period: Period 2
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 86 | 97
Completed | 77 | 87
Not Completed | 9 | 10
Not completed — Death | 0 | 1
Not completed — AE Related to Study Drug | 0 | 1
Not completed — AE not Related to Study Drug | 4 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Reason not Specified | 0 | 2
Period: Follow-up
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 77 | 87
Completed | 77 | 86
Not Completed | 0 | 1
Not completed — AE not Related to Study Drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Pregabalin: Participants were randomized to double-blind treatment with placebo for 6 weeks in period 1 followed by pregabalin in period 2 (2 week dose titration [starting dose: 150 mg/day] and 4 weeks fixed dose [150 - 300 mg/day]). There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
- Total: Total of all reporting groups
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (8.5) | 58.4 (9.3) | 58.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 61 | 71 | 132

OUTCOME MEASURES:

1. Primary Outcome: Average Diabetic Peripheral Neuropathy (DPN) Pain Based on a Numeric Rating Scale (NRS) Over the Last 7 Days of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The daily pain diary consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by having chosen the appropriate number between 0 and 10. Self-assessment was performed daily each evening before bedtime (6.00 pm to midnight) on the telephone via Interactive Voice Recognition System (IVRS). The endpoint mean pain score was defined as the mean of the last 7 daily diary pain ratings while taking study medication in each treatment period - Period 1 and Period 2, respectively. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: All participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation were included in the Intent-to-Treat (ITT) analysis (N: 203). This was the primary analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Pregabalin: The below table included data from participants while receiving pregabalin in either period of the 2-period crossover study design. This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (2 weeks dose titration and 4 weeks fixed dose for each treatment period). There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
- Placebo: The below table included data from participants while receiving placebo in either period of the 2-period crossover study design. This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (2 weeks dose titration and 4 weeks fixed dose for each treatment period). There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 4.73 (0.14) | 4.96 (0.14)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model including baseline pain, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. Last observation carried forward (LOCF) approach was applied; Test type: Superiority or Other; p = 0.0659, Linear mixed effects model — Primary analysis was two-sided and performed at the 0.05 significance level. The study was considered positive only if both co-primary endpoints had p-values that were less than 0.05, hence there was no need for multiplicity adjustment; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.46 to 0.01], Standard Error of Mean 0.12

2. Post Hoc Outcome: Average Weekly DPN Pain Based on a NRS (Baseline, 6 Weeks in Period 1, 2 Weeks Washout and 6 Weeks in Period 2)
Description: The daily pain diary consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by having chosen the appropriate number between 0 and 10. Self-assessment was performed daily each evening before bedtime (6.00 pm to midnight) on the telephone via IVRS. The longitudinal mean weekly DPN pain scores were defined as the mean of 7 daily diary pain ratings. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: Baseline, 6 weeks in Period 1, 2 weeks washout and 6 weeks in Period 2
Population: All participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation were included in the ITT analysis (N: 203). Numbers of participants analyzed are provided in section Measured Values in brackets (N: Pregabalin, Placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale
  V6 (N: 101, 102) | 4.66 (1.77) | 5.29 (1.93)
  V11 (N: 97, 84) | 4.57 (2.22) | 4.38 (2.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; This longitudinal analysis was a sensitivity analysis of the primary endpoint. P-value was based on a repeated measure mixed effects model including pooled center, time point, treatment, an indicator variable for Week 6 as well as interaction terms as fixed effect factors. For analysis purpose, it is assumed that participants were on placebo at Baseline, took the same treatment as in Period 1 during Week 1 of washout, and were on placebo in Week 2 of washout; Test type: Superiority or Other; p = 0.0242, Repeated measure mixed effects model — Primary analysis was two-sided and performed at the 0.05 significance level. Unstructured covariance structure was used to estimate the within-participant errors; The Kenward-Roger method was used to estimate denominator degrees of freedom; Mean Difference (Final Values) = -0.291, 95% CI 2-sided [-0.543 to -0.038], Standard Error of Mean 0.128

3. Primary Outcome: DPN Pain on Walking Based on a 11-point NRS of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The post-test DPN pain on walking NRS consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their DPN pain in their legs and/or feet while walking during the 50-foot walk test by choosing the appropriate number between 0 and 10. The post-test DPN pain on walking NRS was completed by the participant using paper-pen administration immediately after completing the 50-foot walk test at the end of each treatment period - Period 1 and Period 2, respectively. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: All participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation were included in the ITT analysis (N: 203). This was the primary analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 4.28 (0.15) | 4.41 (0.15)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a repeated measure linear mixed effects model including baseline pain, sequence, period, center, time, treatment, and treatment by time interaction as fixed effect factors and participant within sequence and within-participant error as random factors. The model term 'time' may take 2 values corresponding to Week 3 and Week 6 in each period; Test type: Superiority or Other; p = 0.4120, Mixed-Effect Model Repeated Measures — Primary analysis was two-sided and performed at the 0.05 significance level. The study was considered positive only if both co-primary endpoints have p-values that are less than 0.05, hence there was no need for multiplicity adjustment; Satterthwaite's approximation was used to estimate denominator degrees of freedom; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.44 to 0.18], Standard Error of Mean 0.16

4. Secondary Outcome: Percentage of Participants Achieving 30% Reduction in Mean DPN Pain Score From Baseline at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The daily pain diary consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by having chosen the appropriate number between 0 and 10. Self-assessment was performed daily each evening before bedtime (6.00 pm to midnight) on the telephone via IVRS. The endpoint mean pain score was defined as the mean of the last 7 daily diary pain ratings while taking study medication in each treatment period - Period 1 and Period 2, respectively. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: All participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation were included in the ITT analysis (N: 203). This was the primary analysis set. Numbers of participants analyzed are provided in section Measured Values in brackets (N: Pregabalin, Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
percentage of participants
  V6 (N: 101, 102) | 38.6 | 24.5
  V11 (N: 97, 84) | 46.4 | 47.6
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done overall (period 1 and period 2) using a generalized linear mixed model which included response as the dependent variable, sequence, period, pooled center, treatment as fixed effects, and subject within treatment as random effect. LOCF approach was applied; Test type: Superiority or Other; p = 0.0847, Generalized linear mixed model — Secondary analysis was two-sided and performed at the 0.05 significance level. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.94 to 2.55]

5. Secondary Outcome: Percentage of Participants Achieving 50% Reduction in Mean DPN Pain Score From Baseline at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 4
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
percentage of participants
  V6 (N: 101, 102) | 23.8 | 13.7
  V11 (N: 97, 84) | 27.8 | 32.1
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2459, Generalized linear mixed model — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.80 to 2.39]

6. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) Score for Pain-Severity Domain at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. The BPI-sf consists of 5 questions: 4 items measure pain (0: no pain; 10: worst pain possible) at its "worst, "least", "average", and "now" (current pain) on an 11-point scale. Scores range from 0 - 40 with higher scores indicating greater pain severity. Another item, containing 7 sub-questions, evaluates the level of interference of pain on daily functioning (general activity, walking, work ability, mood, enjoyment of life, relations with other people, and sleep) on 11-point scales (0: does not interfere; 10: completely interferes). Scores range from 0 - 70 with higher scores indicating greater interference.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 16.76 (0.56) | 17.56 (0.75)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model including baseline pain, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0889, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.71 to 0.12], Standard Error of Mean 0.46

7. Secondary Outcome: BPI-sf Score for Pain-Interference Domain at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 6
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 22.58 (0.96) | 23.75 (0.98)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1781, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.86 to 0.53], Standard Error of Mean 0.86

8. Secondary Outcome: BPI-sf Score for Pain-Interference With Walking Ability at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. The BPI-sf consists of 5 questions: 4 items measure pain on an 11-point scale. Scores range from 0 - 40 with higher scores indicating greater pain severity. Another item, containing 7 sub-questions, evaluates the level of interference of pain on daily functioning (general activity, walking, work ability, mood, enjoyment of life, relations with other people, and sleep) on 11-point scales (0: does not interfere; 10: completely interferes). Scores range from 0 - 70 with higher scores indicating greater interference. The sub-score pain interference with walking ability was evaluated, as it was considered to be the most relevant in the context of this study.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 3.75 (0.17) | 3.93 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.2719, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.53 to 0.15], Standard Error of Mean 0.17

9. Secondary Outcome: Daytime Total Activity Counts Per Day Measured by Actigraphy Over the Last 7 Days of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Actigraphy data which measured steps and daytime activity during waking hours were assessed for the last 7 days at Baseline, Visit 6, and Visit 11. Activity counts are the units of motion. It is equal to the sum of peak accelerations each second during the epoch (60 seconds). Total activity counts per day is the sum of the activity counts for each epoch (60 seconds) during the "day" (non-sleep period). Actigraphy was performed with an accelerometer that was worn on the hip during the waking hours. It was programmed to record movements while the device was being worn.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: counts
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
counts | 64703.14 (4005.00) | 64139.75 (4057.89)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model including baseline value, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. LOCF approach was applied; Test type: Superiority or Other; p = 0.8909, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 563.39, 95% CI 2-sided [-7549.82 to 8676.60], Standard Error of Mean 4098.74

10. Secondary Outcome: Steps Per Day Measured by Actigraphy Over the Last 7 Days of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Actigraphy data which measured steps and daytime activity during waking hours were assessed for the last 7 days at Baseline, Visit 6, and Visit 11. The participants were instructed to wear the device on their hip during the waking hours.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: steps
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
steps | 3785.65 (201.17) | 3788.28 (203.05)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.9899, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-411.26 to 406.01], Standard Error of Mean 206.37

11. Secondary Outcome: Walk 12 Questionnaire Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The Walk-12 is a self-administered questionnaire that assesses the impact of the participant's diabetic neuropathy over the past 2 weeks on parameters associated with walking (12 questions) based on a 5-point scale (from not at all to extremely). The total score is the sum of scores from the 12 questions, which then gets transferred to a 0-100 scale with higher scores indicating greater impairment
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 35.72 (1.44) | 37.08 (1.46)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model including baseline value, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.2854, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-3.88 to 1.15], Standard Error of Mean 1.27

12. Secondary Outcome: Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QOL-DN) Total Quality of Life (TQOL) Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. TQOL score should be summed as follow: sum (Σ) (1 - 7, 8 - 35). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 29.31 (1.17) | 30.77 (1.19)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1805, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-3.60 to 0.68], Standard Error of Mean 1.09

13. Secondary Outcome: Norfolk QOL-DN Symptoms Domain Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. The symptoms domain score should be summed as follow: Σ(1 - 7, 9). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 7.65 (0.32) | 7.99 (0.33)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.3028, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.99 to 0.31], Standard Error of Mean 0.33

14. Secondary Outcome: Norfolk QOL-DN Activities of Daily Living Domain Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. The activities of daily living domain score should be summed as follow: Σ(12, 22, 23, 25, 26). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 2.36 (0.19) | 2.42 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.7542, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.41 to 0.30], Standard Error of Mean 0.18

15. Secondary Outcome: Norfolk QOL-DN Physical Functioning / Large Fiber Domain Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. The physical functioning / large fiber domain score should be summed as follow: Σ(8, 11, 13 - 15, 24, 27 - 35). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 15.51 (0.73) | 16.78 (0.75)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0634, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.62 to 0.07], Standard Error of Mean 0.68

16. Secondary Outcome: Norfolk QOL-DN Small Fiber Domain Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. The small fiber domain score should be summed as follow: Σ(10, 16, 17, 18). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 2.77 (0.17) | 2.53 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1985, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.13 to 0.62], Standard Error of Mean 0.19

17. Secondary Outcome: Norfolk QOL-DN Autonomic Domain Score Measured Over the Last 2 Weeks of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With the exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. The autonomic domain score should be summed as follow: Σ(19, 20, 21). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 1.07 (0.10) | 1.08 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.9686, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.21 to 0.20], Standard Error of Mean 0.10

18. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGIC) Score From Baseline at the End of Period 1 (Week 6)
Description: The PGIC is a participant-rated instrument that measures the participant's assessment of change in his/her overall status on a scale ranging from 1 (very much improved) to 7 (very much worse). Original scores (OS; 7 different scores) and categorized scores (CS; 4 different scores) were provided. Categorized scores were very much improved (consisting of very much improved and much improved); any improvement (consisting of very much improved, much improved, and minimally improved); no change (consisting of no change); and any worsening (consisting of minimally worse, much worse, and very much worse). Due to the crossover design, PGIC was analyzed at the end of period 1 (V6).
Time Frame: End of Period 1 (V6)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 98 | 102
percentage of participants
  OS: Very much improved | 11.2 | 5.9
  OS: Much improved | 39.8 | 25.5
  OS: Minimally improved | 30.6 | 27.5
  OS: No change | 13.3 | 33.3
  OS: Minimally worse | 2.0 | 5.9
  OS: Much worse | 2.0 | 1.0
  OS: Very much worse | 1.0 | 1.0
  CS: Very much improved | 51.0 | 31.4
  CS: Any improvement | 81.6 | 58.8
  CS: No change | 13.3 | 33.3
  CS: Any worsening | 5.1 | 7.8
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Odds ratio is based on the binary response for any improvement while p-value is from the comparison of the original scale of 7 possible outcomes. P-value was calculated by using Cochran Mantel-Haenszel (CMH) test. PGIC values at the end of Period 1 data was compared between treatment groups; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.5400, 95% CI 2-sided [1.30 to 4.95]

19. Secondary Outcome: Mean Sleep Interference Rating Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The daily sleep diary consists of an 11-point numeric rating scale with which the participant rates how painful DPN pain has interfered with their sleep during the past 24 hours. Zero indicates "does not interfere with sleep" and 10 indicates "completely interferes (unable to sleep due to pain)". Self-assessment was performed daily in the evening before bedtime on a telephone via IVRS (time window for completion between 6.00 pm to midnight) after completion of the daily pain diary.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 3.66 (0.12) | 4.05 (0.13)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0105, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.68 to -0.09], Standard Error of Mean 0.15

20. Secondary Outcome: Hospital Anxiety and Depression Scale - Anxiety (HADS-A) Total Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale consists of 7 statements and the participant responds as to how each item applies to him/her over the past week on 4-point response scale. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 4.65 (0.19) | 4.92 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1178, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.63 to 0.07], Standard Error of Mean 0.18

21. Secondary Outcome: Hospital Anxiety and Depression Scale - Depression (HADS-D) Total Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The HADS is a 14-item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale consists of 7 statements and the participant responds as to how each item applies to him/her over the past week on 4-point response scale. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale | 3.73 (0.20) | 3.97 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1990, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.60 to 0.13], Standard Error of Mean 0.18

22. Secondary Outcome: Euro QoL-5 Dimensions (EQ-5D) - Health State Profile Utility Scores at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The EQ-5D describes participant's health status based on 5 attributes producing an 5 digit index score. The 5 dimensions are: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Dolan 1997 advised how to transfer this index score to a single score for clinical trials, a revised single index was published in 2001. The index uses general population weighted estimates for various health states. In general, the range of the single index tends to vary between 0 = death and 1 = perfect health and there are some states that have been rated by the general population to be worse than death which may result in numbers below 0.
Time Frame: End of Period (includes both Visits 6 and 11)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 198 | 186
units on a scale
  Index score Dolan 1997 | 0.649 (0.015) | 0.643 (0.015)
  Index score Dolan 2001 | 0.650 (0.014) | 0.641 (0.014)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the Index score Dolan 1997. Analysis was done using a linear mixed effects model including baseline value, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.71107, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.025 to 0.037], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the Index score Dolan 2001. Analysis was done using a linear mixed effects model including baseline value, sequence, period, center, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.53965, Linear mixed effects model — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.009, 95% CI 2-sided [-0.021 to 0.039], Standard Error of Mean 0.02

ADVERSE EVENTS:
Time Frame: From the time that the participants were provided the informed consent document through and including 28 calendar days after the last administration of the study drug.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 9/198 | 2/186
Other Adverse Events (participants affected / at risk) | 53/198 | 38/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=198) | Placebo (N=186)
Angina unstable (Cardiac disorders) | 1 | 0
Myocardial infarction (Endocrine disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0 — The participant received pregabalin in period 2, when he/she experienced the SAE of drug withdrawal convulsions.
Fracture treatment (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=198) | Placebo (N=186)
Vision blurred (Eye disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 6
Fatigue (General disorders) | 11 | 3
Oedema peripheral (General disorders) | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Weight increased (Investigations) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Dizziness (Nervous system disorders) | 11 | 6
Headache (Nervous system disorders) | 5 | 8
Somnolence (Nervous system disorders) | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.